CLINICAL TRIAL: NCT01033513
Title: SOS Nutrition Project
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Charlotte (Other)
Collaborators: Administration on Aging, United States (U.S. Federal Agency); Mecklenburg County Department of Social Services (Unknown)
Responsible Party: William J. McAuley
Other Study IDs: AoA90AM2665
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Literature Only (Control): The participants on this arm served as the control group. Five types of literature were mailed to the participants in the literature only arm. A letter was included with the materials thanking participants for their participation, requesting that the participants read the literature, and encouraging them to contact the RDs with any questions. The Clinical Study Manager's telephone number was provided for questions about diet or lifestyle changes. The RDs documented all contacts with participants on a phone summary. Other than the delivery of literature and responses to specific questions asked by the participant or the participant's primary caregiver through telephone calls, the RDs had no further interaction with the participant until the conclusion of the participant's trial period.
- Meals Only: Participants in the meals only arm received a pre-intervention assessment (but no nutrition counseling). The RDs gave the participants in the meals only arm a phone number and encouraged them to phone with questions or problems, especially problems associated with the meals. Subsequently, the meals only participants received seven diagnosis-appropriate therapeutic meals a week, delivered once per week. The meals were specially designed to address the participants' medical diagnoses. They were developed using the ADA MNT protocols for caloric and nutrient content requirements for individuals with the specified diagnoses, in addition to meeting AoA Nutrition Program dietary requirements. The meals were provided primarily in frozen form. However, some shelf-stable and refrigerated components were also included. In conformance with AoA regulations, appropriate meals were also offered to the spouse of any participant receiving a therapeutic meal.
- MNT Only: The participants in this arm received MNT from the project RDs, who employed the Hyperlipidemia Medical Nutrition Therapy MNT Protocol, developed by ADA (2002). Because ADA had not finalized MNT protocols for hypertension, the RDs followed the protocol for hyperlipidemia for participants diagnosed with either hyperlipidemia or hypertension, with adjustments, as appropriate, to benefit those individuals who were diagnosed with hypertension.All MNT sessions were in the participants' homes, and if a caregiver was required for the individual to participate in the project, every effort was made to include this person in the MNT sessions. The MNT intervention took place over at least three sessions, and, in conformance with the ADA protocol, each participant received individualized counseling and education.
- Meals and MNT: The participants assigned to the MNT plus meals arm received both of the interventions, as described above.

SUMMARY:
Many older people experience hyperlipidemia and hypertension, but, to date, there is little information regarding whether or not medical nutrition therapy (MNT) or therapeutic meals have an independent or joint beneficial impact on older people with these diagnoses. This report describes a clinical trial in which the investigators directly examined these issues. Two key clinical outcome measures include changes in diastolic blood pressure and total fasting serum cholesterol. In addition to these clinical outcome measures the investigators collected health related quality of life data and data that permitted cost-effectiveness analyses.

The investigators hypothesized that MNT and therapeutic meals would each lead to lower total fasting serum cholesterol and lower diastolic blood pressure after the 52-week trial, in comparison to individuals who received standard support (commonly available literature on how to manage their disease). The investigators also hypothesized that MNT plus therapeutic meals would be especially beneficial because of their synergistic effects on the clinical outcomes. Although the investigators established no specific hypotheses regarding the potential impact of MNT or therapeutic meals on cost of care and quality adjusted life years, the investigators were interested in whether MNT or therapeutic meals would be associated with these two measures.

ELIGIBILITY:
Inclusion Criteria:

* People were eligible for the study if they were 60 years old or older and: *were diagnosed by a physician with hyperlipidemia and/or hypertension

  * had storage space for frozen and shelf-stable meals
  * had the mental and physical capacity to safely store, prepare, and consume meals and benefit from MNT
  * had their physician's permission to be included in the trial
  * were willing/able to provide blood samples, stay on the regimen, maintain the healthcare/medication utilization diary, and answer questions about diet and quality of life
  * were willing to stay on the their arm and consume meals and/or receive MNT if assigned to one of those arms
  * did not leave their town or city in a typical week unless it was for reasons that are acceptable under the Medicare definition of homebound
  * did not plan to be away from home for more than two weeks during the intervention period
  * were able to communicate (speak, read, write) in English and were able to understand and willing to complete the consent process for participation.

Exclusion Criteria:

* Individuals excluded from the study were those younger than age 60, or those without one of the qualifying diagnoses (hypertension or hyperlipidemia), and those who had any of the following characteristics:

  * coronary artery bypass, diabetes, myocardial infarction within the 12 months prior to enrollment, renal insufficiency, major surgery in the 12 weeks prior to enrollment, unstable angina, uncompensated congestive heart failure, liver disease, pancreatic disease, current serious gastrointestinal disease (for example, colitis), or current cancer or other life-limiting diagnoses
  * were unable to safely manage and consume frozen and shelf stable meals
  * self-disclosed as having alcohol or drug abuse within the 24 months prior to enrollment
  * were unable or unwilling to provide necessary biological material and other information required by the study
  * had very high knowledge of dietary/lifestyle management issues required by the diagnosis, based on a knowledge questionnaire
  * indicated that they left their city or town in a typical week
  * were employed full-time
  * had significant food allergies or were unable to eat the food offered through the project because of religious or other restrictions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See inclusion and exclusion criteria below.
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2003-05; Study Completion 2006-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J McAuley, PhD, Principal Investigator — George Mason University